CLINICAL TRIAL: NCT05251402
Title: The ALOHA Trial: Addressing Quality of Life, Clinical Outcomes, and Mechanisms in Uncontrolled Asthma Following the DASH Dietary Pattern
Brief Title: Addressing Quality of Life, Clinical Outcomes, and Mechanisms in Uncontrolled Asthma Following the DASH Dietary Pattern
Acronym: ALOHA
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Stanford University (Other); University of Vermont (Other); University of Newcastle, Australia (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Chicago (Other)
Responsible Party: Principal Investigator, Jun Ma, Beth and George Vitoux Professor of Medicine, Department of Medicine, Principal Investigator, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-1375; R61HL155160 (NIH)
Record Dates: First submitted 2022-02-02; First posted 2022-02-22 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Patinet Education (Active Comparator): If you are assigned to this group, you will receive education on asthma and health from an ALOHA health coach.
  Interventions: Behavioral: Group A - Patient Education
- Group B - Patient Education with Nutrition Counseling (Active Comparator): If you are assigned to this group, you will receive the same patient education on asthma and health as Group A. In addition, you will receive nutrition counseling from your health coach who is a registered dietitian.
  Interventions: Behavioral: Group B - Patient Education with Nutrition Counseling

INTERVENTIONS:
Behavioral: Group A - Patient Education — If you are assigned to this group, you will receive education on asthma and health from an ALOHA health coach.
  * In months 1-3, you will attend 3 individual and 8 group sessions. Individual sessions will last ~15 minutes and the first one will be in-person. Group sessions will last ~30 minutes and the first 2 of the 8 will be in person. You and your coach will determine if you may attend the remaining individual and group sessions remotely instead, via Zoom or phone. The purpose of these sessions is to provide you with general information about respiratory health topics, including recommendations for asthma care, inhaler use, and lung health.
  * In months 4-12, you will complete 11 phone check-ins for ~10 minutes each. The purpose of these phone calls is to provide you with ongoing support and discuss health topics of your choice.
  Arms: Group A - Patinet Education
Behavioral: Group B - Patient Education with Nutrition Counseling — If you are assigned to this group, you will receive the same patient education as Group A. In addition, you will receive nutrition counseling from your health coach who is a registered dietitian.
  * In months 1-3, the duration of the sessions will increase to ~30 minutes each for the 3 individual sessions and to ~60 minutes each for the 8 group sessions. This is because in addition to providing the same information on asthma and health as in Group A, your health coach will also counsel you on how to follow the DASH diet by adopting effective behavior change techniques such as goal setting, self-monitoring, and problem solving.
  * In months 4-12, your health coach will review your progress, provide you with personalized feedback, assist you in problem solving as you continue to work towards the DASH dietary goals, and help you maintain the changes you have made over the long term.
  Arms: Group B - Patient Education with Nutrition Counseling

SUMMARY:
The goal of the ALOHA trial is to investigate the efficacy of improved diet quality following a DASH behavioral intervention that has shown promising results in adults with uncontrolled asthma. DASH stands for Dietary Approaches to Stop Hypertension. This healthy diet is known to help people with high blood pressure manage their health. But physicians do not know if the DASH diet can also benefit patients with uncontrolled asthma. Researchers in the ALOHA study are trying to find out the answer to this important question.

Researchers at UIC are studying how 2 asthma care programs compare in terms of helping adults with uncontrolled asthma to improve their quality of life. Researchers also want to learn what might explain the differences in patient outcomes that they may see between the 2 programs.

The primary outcome will be asthma-specific quality of life. If the DASH behavioral intervention is found to benefit people with uncontrolled asthma, it would provide a practical, safe, and acceptable public-health intervention in the form of dietary modification to reduce the burden of asthma.

DETAILED DESCRIPTION:
Approximately 320 subjects who are determined fully eligible will be randomly assigned (by chance, like flipping a coin) to participate in intervention Group A or Group B, where you will receive either 1 of the 2 asthma care programs

Both asthma care programs are for a year and offer patient education on asthma and health. In both asthma care programs, you will receive fact-based patient information on asthma and health. Additionally, in one of the programs, a registered dietitian will also provide nutrition counseling on how to follow the USDA recommended DASH diet. Both asthma care programs offer 3 individual sessions, 8 group sessions, and 11 phone consultations. Your first individual session will be in-person with a trained health coach on the ALOHA team. The remaining 2 individual sessions will be either in-person or remote, depending on what you and your coach decide. You will also attend the first 2 (of 8) group sessions in-person to build connection with your coach and peer participants in the group. You and your coach will then decide whether you should attend the remaining group sessions in-person or remotely. Your ALOHA health coach will offer you continued support by phone until you complete your 1-year program.

Study Visits at UIC: Irrespective of your asthma care group, all participants will be expected to visit UIC Study site 4 times over the next year, initially and then at 3 months, at 6 months, and finally at one year. You will meet with an ALOHA study coordinator for 2 hours at the initial and final visits and for 1 hour at 3 and 6 months. Before each visit, you will complete online surveys about your health and phone interviews about your diet. At each visit, you will complete a breathing test, a blood draw, a physical exam, and questions about your asthma, diet and exercise habits, use of asthma medications and dietary supplements.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at study enrollment
* Diagnosis of asthma with currently prescribed controller therapy (i.e., Step 2 or above) according to the 2020 asthma guideline update (EPR4)
* Uncontrolled asthma on study screening based on Asthma Control Test (ACT) scores <20
* Being able and willing to provide written informed consent and HIPAA authorization

Exclusion Criteria:

* Inability to speak, read or understand English sufficiently to provide valid informed consent
* Primary diagnosis of COPD (emphysema or chronic bronchitis)
* Previous cardiovascular disease: coronary heart disease (myocardial infarction, angina pectoris, percutaneous coronary intervention, coronary artery bypass graft surgery), cerebrovascular disease (stroke, transient ischemic attack), peripheral vascular disease, heart failure, or aortic aneurysm
* Diabetes (other than during pregnancy)
* Diagnosis of cancer (other than non-melanoma skin cancer) within the past year and/or actively receiving cancer treatment
* Inflammatory bowel disease, colostomy, malabsorption, or major gastrointestinal resection
* Diagnosis of bipolar or psychotic disorder
* Hospitalization for psychological or emotional problems within the last 2 years
* Cognitive impairment based on the Callahan 6-item screener67
* Terminal illness or in hospice or long-term care
* Current diet of good quality (DASH concordance index ≥6 out of 9 total)
* Current/planned participation in another structured program that overtly focuses on diet and nutrition
* On special diet that precludes changes adherent to the DASH dietary pattern or otherwise unwillingness to modify current diet
* Current use of prescription or non-prescription weight-loss products and unwillingness to stop taking them for the duration of the study
* Underweight per body mass index (BMI) below 18.5 kg/m2 based on measured height and weight at study enrollment
* Actively attempting to lose weight or weight change >15 lbs during prior 3 months
* Active alcohol or substance use disorder (including prescription drugs) based on the CAGE Questionnaire Adapted to Include Drugs (CAGE-AID)68
* Current within the past 6-months or former smoker (more than 20-packs of cigarettes in the lifetime, or current smoker)
* Current or planned pregnancy or currently lactating
* Planning to move out of the area during the study period
* Participation in another clinical trial or investigational treatment study
* Family/household member of an already enrolled participant or of a study team member
* Investigator discretion for clinical safety or protocol adherence reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving a clinically significant improvement (responders) in asthma-specific quality of life (Aim 1) | Baseline, 3 months, 6 months, 12 months
  The 15-item Juniper Mini Asthma-Specific Quality of Life Questionnaire (AQLQ) has been shown to have excellent reliability and responsiveness to change in asthma control. It consists of 5 items on symptoms, 4 items on activity limitations, 3 items on emotional function, and 3 items concerning environmental stimuli. Each item is rated on a scale from 1=maximum impairment to 7=no impairment over the last 2 weeks. The overall AQLQ score is an average of the item scores equally weighted. The primary outcome is the percentage of participants achieving the minimal clinically important difference (MCID) of at least a 0.5-point increase in AQLQ scores from baseline to 12 months. The percentages of responders at 3 and 6 months are secondary outcomes.

SECONDARY OUTCOMES:
Level of asthma-specific quality of life (Aim 1) | Baseline, 3 months, 6 months, 12 months
  The overall AQLQ score is the mean of all the items on the Mini AQLQ. Items are equally weighted. A domain score is calculated as the mean of all the items within each of the 4 domains: symptoms, activity limitations, emotional function, and environmental stimuli. Changes in overall and domain scores from baseline to each follow-up time point are secondary outcomes.
Level of asthma control (Aim 1) | Baseline, 3 months, 6 months, 12 months
  The overall ACQ score is an average of the item scores equally weighted and ranges from 0=well controlled to 6=extremely poorly controlled. Change in ACQ scores from baseline to each follow-up time point are secondary outcomes.
Proportion of participants achieving a clinically significant improvement (responders) in asthma control (Aim 1) | Baseline, 3 months, 6 months, 12 months
  The Juniper Asthma Control Questionnaire (ACQ) is a validated composite measure of asthma control recommended for research purposes. It consists of 7 items on daytime and nocturnal symptoms, activity limitations, rescue medication use (excluding prophylactic use for exercise-induced bronchospasm), and FEV1% of predicted norm. Each item is rated on a 7-point scale from 0 (least severe) to 6 (most severe). ACQ has been validated for self-administration (except for the FEV1 item, which is obtained by spirometry) and has high internal reliability (intra-class correlation coefficient=0.90). The overall ACQ score is an average of the item scores equally weighted. The proportion of responders is the percentage of participants achieving the MCID of at least a 0.5-point increase in ACQ scores. Percentages at each follow-up time point are secondary outcomes.
Level of Pre-bronchodilator measurements of FEV1 (Aim 1) | Baseline, 3 months, 6 months, 12 months
  Lung function will be assessed by forced spirometry as per the American Thoracic Society (ATS) standards, both before and after bronchodilator. Post-bronchodilator spirometry will be performed at 15 minutes and 2 hours after bronchodilator administration. Participants will be instructed to refrain from taking inhaled medications for breathing during the 6-24 hours prior to their visit depending on the medication, unless they are having trouble with their breathing. Participants will blow forcefully for at least 6 seconds for 3-8 times until 3 acceptable results show repeatability. Spirometry outcomes for Aim 1 include PRE-bronchodilator measurements of forced expiratory volume in 1 second (FEV1)
Level of Pre-bronchodilator measurement of FVC (Aim 1) | Baseline, 3 months, 6 months, 12 months
  Lung function will be assessed by forced spirometry as per the American Thoracic Society (ATS) standards, both before and after bronchodilator. Post-bronchodilator spirometry will be performed at 15 minutes and 2 hours after bronchodilator administration. Participants will be instructed to refrain from taking inhaled medications for breathing during the 6-24 hours prior to their visit depending on the medication, unless they are having trouble with their breathing. Participants will blow forcefully for at least 6 seconds for 3-8 times until 3 acceptable results show repeatability. Spirometry outcomes for Aim 1 include PRE-bronchodilator measurements of forced vial capacity (FVC).
Level of Pre-bronchodilator measurements FEV1/FVC (Aim 1) | Baseline, 3 months, 6 months, 12 months
  Lung function will be assessed by forced spirometry as per the American Thoracic Society (ATS) standards, both before and after bronchodilator. Post-bronchodilator spirometry will be performed at 15 minutes and 2 hours after bronchodilator administration. Participants will be instructed to refrain from taking inhaled medications for breathing during the 6-24 hours prior to their visit depending on the medication, unless they are having trouble with their breathing. Participants will blow forcefully for at least 6 seconds for 3-8 times until 3 acceptable results show repeatability. Spirometry outcomes for Aim 1 include PRE-bronchodilator measurements of FEV1/FVC.
Level of asthma medication adherence (Aim 1) | Baseline, 3 months, 6 months, 12 months
  The Adult Asthma Adherence Questionnaire is a validated and practical questionnaire that reflects nonadherence risk and identifies potential adherence barriers.
Count of episodes of poorly controlled asthma (Aim 1) | Baseline, 3 months, 6 months, 12 months
  Episodes of poorly controlled asthma will be assessed as per a modified ALA-ACRC definition if any of the following apply: (1) addition of oral corticosteroid (prednisone or prednisolone) to treat asthma symptoms or (2) unscheduled contact with a health care provider (ED visit, physician office, hospital) for asthma symptoms.
Measure overall health-related quality of life | Baseline, 3 months, 6 months, 12 months
  The 12-item Short-Form Health Survey (SF-12) is a 12-item version of the SF-36 that measures overall health-related quality of life. Physical and mental health composite scores are computed using the scores of 12 questions and range from 0 to 100, with 0 indicating the lowest level of health and 100 indicating the highest level of health. Test-retest correlation is 0.89 for the physical health subscale and 0.76 for the mental health subscale.
Level of Blood pressure (BP) (Aim 1) | Baseline, 3 months, 6 months, 12 months
  The American Heart Association recommendations for BP measurement will be followed. Participants will be told not to engage in vigorous exercise, ingest food or caffeine, or smoke within a half hour of BP measurements. If a half hour has not elapsed, the BP measurements must be delayed until a half hour has passed. BP will be measured in the seated position after at least a 5-minute rest in a quiet room where no other activity is taking place and where temperature fluctuations are minimal. At baseline, both arms will be measured once and 2 more times on the arm with higher systolic reading using standard equipment at participating clinics. This same arm will be measured 3 times at each follow-up assessment. Wait 1 minute between each measurement.
Level of psychological distress (Aim 1) | Baseline, 3 months, 6 months, 12 months
  The Depression, Anxiety and Stress Scale-21 items (DASS21) is a set of 3 self-report scales designed to measure the emotional states of depression, anxiety, and stress. Each of the 3 scales contains 7 items. Each item is scaled from 0 (did not apply to me at all) to 3 (applied to me very much or most of the time). The depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest/involvement, anhedonia and inertia. The anxiety scale assesses autonomic arousal, skeletal muscle effects, situational anxiety, and subjective experience of anxious affect. The stress scale assesses difficulty relaxing, nervous arousal, and being easily upset/agitated, irritable/over-reactive and impatient. Each scale is scored as the sum of the item scores.
Level of sleep disturbance (Aim 1) | Baseline, 3 months, 6 months, 12 months
  Sleep quality will be assessed on the 8-item PROMIS sleep disturbance (SD) scale. It measures symptoms of insomnia. Each item is scaled from 1 (not at all) to 5 (very much).
Level of sleep-related impairment (Aim 1) | Baseline, 3 months, 6 months, 12 months
  The 8-item PROMIS sleep-related impairment (SRI) scale measures symptoms of daytime sleepiness. Each item is scaled from 1 (not at all) to 5 (very much). Correlation between the SD short form and the Pittsburgh Sleep Quality Index (PSQI, hypothesized to measure similar attributes) is 0.83 and correlation between the SRI short form and the Epworth Sleepiness Scale (ESS, hypothesized to measure a related but slightly different construct, the propensity to doze during activities) is 0.46, similar to the correlations between the SD full banks and PSQI (0.85) and between SRI full banks and the ESS (0.45).
Degree of bronchodilator responsiveness based on pre- and post-bronchodilator percent change in FEV1 (Aim 2) | Baseline, 3 months, 6 months, 12 months
  Bronchodilator responsiveness will be measured based on percent change in FEV1 from prebronchodilator to 15 minutes and 2 hours postbronchodilator. Forced spirometry will be performed as per the American Thoracic Society (ATS) standards both before and after bronchodilator. Post-bronchodilator spirometry will be performed at 15 minutes and 2 hours after bronchodilator administration. Participants will be instructed to refrain from taking inhaled medications for breathing during the 6-24 hours prior to their visit depending on the medication, unless they are having trouble with their breathing. Participants will blow forcefully for at least 6 seconds for 3-8 times until 3 acceptable results show repeatability.
Level of plasma short chain fatty acids (propionate, butyrate, and acetate) (Aim 2) | Baseline, 3 months
  Circulating short chain fatty acids (SCFA) will be measured with approximately 4 cc serum, aliquoted into 200 µl cryovials and kept frozen at -80°C. These samples will be shipped overnight on dry ice to the University of Michigan metabolomic core for measurement of propionate, butyrate and acetate, as circulating measures of products of gut microbial fermentation.
Level of PBMC cytokines (Interferon-γ, IL-5, IL-17A, IL-10, IL-1β, IL-6, IL-8, TNFα) (Aim 2) | Baseline, 3 months
  To measure changes in adaptive and innate immune function pertinent to obese asthma, we will use the Tru-Culture® (myriad RBM tubes, 1 cc blood for each tube): one containing TruCulture® media + 0.1 μg/mL lipopolysaccharide, one containing TruCulture® media + 0.4 μg/mL anti-CD3, and one containing TruCulture® media alone. Samples will be incubated upright in a dry heat block at 37°C for 24 hours. Supernatant and cells will be isolated and frozen at -80°C, then shipped overnight on dry ice to the University of Vermont for cytokine and gene expression studies, respectively. For effects on T cell function pertinent to adaptive immunity we will measure cytokines pertinent to TH1 (interferon gamma), TH2 (IL-5), TH17 (IL-17A) and Tregs (IL-10) in media from cells incubated with anti-CD3 versus media alone. For effects on mononuclear cell responses pertinent to innate immunity, we will measure IL-1β, IL-6, IL-8 and TNFα in response to lipopolysaccharide versus media.
Level of diet quality based DASH score (Aim 3) | Baseline, 3 months, 6 months, 12 months
  Dietary intake will be determined from 3 unannounced 24-hour dietary recalls (2 non-consecutive weekdays and 1 weekend day with a 2-week period) by interview using the US Department of Agriculture multiple pass method. The Nutrition Data System for Research (NDSR) (Minneapolis, MN) will be used for data collection and nutrient analysis. The DASH score using the National Health and Nutrition Survey (NHANES) method sums an individual's adherence points for 9 nutrients (total fat, saturated fat, protein, cholesterol, fiber, magnesium, calcium, sodium and potassium) based on the DASH diet plan. NDSR outputs will provide the values of these 9 nutrients.
Level of diet quality based on the dietary inflammatory index (DII) (Aim 3) | Baseline, 3 months, 6 months, 12 months
  The DII will be applied to dietary intake data collected using the 3 unannounced 24-hour dietary recalls. The DII is a scale developed using data from epidemiologic, animal and in-vitro studies and is a useful marker of diet quality as it quantifies the overall inflammatory potential of diet, which is calculated based on the known inflammatory effects of up to 45 component nutrients and foods.
Level of plasma carotenoids (Aim 3) | Baseline, 3 months, 6 months, 12 months
  4mL blood will be collected in an EDTA tube, centrifuged at 4oC, for 10 minutes at 3000g. Plasma will be stored at -80oC until analysis. High-performance liquid chromatography (HPLC) will be used to measure plasma carotenoid concentrations (lycopene, lutein, β-cryptoxanthin, α-carotene and β-carotene), as an objective indicator of fruit and vegetable intake. Carotenoids will be extracted from plasma samples (with canthaxanthin added as an internal standard) with a series of ethyl acetate and hexane washes. Chromatography will be performed on a Hypersil ODS column with a flow rate of 0.3 mL/min, using mobile phase of acetonitrile:dichloromethane:methanol (0.05% ammonium acetate (85:10:5, vol:vol)). Carotenoids will be detected at 470 nm using a photodiode array detector.

OTHER OUTCOMES:
Level of self-efficacy for dietary change | Baseline, 3 months, 6 months, 12 months
  Self-efficacy for dietary change will be measured using the Eating Habits Confidence Survey. The Eating Habits Confidence Survey is a reliable and valid measure of dietary self-efficacy. Cronbach's alpha coefficients ranged from 0.85 to 0.93 for the 5 factors (resisting relapse, reducing calories, reducing salt, reducing fat, and behavioral skills). Test-retest reliabilities ranged from 0.43 to 0.64.
Level of social support for dietary change | Baseline, 3 months, 6 months, 12 months
  Social support for dietary change will be measured using the Social Support and Eating Habits Survey. Cronbach's alpha coefficients ranged from 0.70 to 0.83 for the friend and family social support subscales.
Level of patient activation | Baseline, 3 months, 6 months, 12 months
  The 13-item Patient Activation Measure (PAM) assesses patient's self-reported knowledge, skill, and confidence for self-managing his or her health condition. It demonstrated acceptable internal consistency (Conbrach's alpha = 0.81). The 13-item PAM score accounts for 92% of the variation in the activity measured by the original 22-item PAM. The score is also significantly correlated with general preventive behaviors and disease-specific self-management behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, MD, PhD, Principal Investigator — University of Illinois at Chicago
Locations (2):
- United States (2):
  - Department of Medicine, Chicago, Illinois
  - UIC CCTS Clinical Research Center, Chicago, Illinois

REFERENCES:
- [Derived] Nyenhuis SM, Dixon A, Wood L, Lv N, Wittels N, Ronneberg CR, Xiao L, Dosala S, Marroquin A, Barve A, Harmon W, Poynter M, Parikh A, Camargo CA Jr, Appel L, Ma J. The effects of the DASH dietary pattern on clinical outcomes and quality of life in adults with uncontrolled asthma: Design and methods of the ALOHA Trial. Contemp Clin Trials. 2023 Aug;131:107274. doi: 10.1016/j.cct.2023.107274. Epub 2023 Jun 26. PMID 37380019